CLINICAL TRIAL: NCT02900430
Title: The Incidence of Invasive Aspergillosis in Acute Myeloid Leukemia
Brief Title: Invasives Aspergillosis in Acute Myeloid Leukemia
Acronym: IA-AML
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: IA-AML
Record Dates: First submitted 2016-09-02; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Acute Myeloid Leukemia; Invasive Aspergillosis
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients without antifungal prophylaxis: Patients with acute myeloid leukemia treated with intensive chemotherapy. From 2009 to 2011, any patient received antifungal (anti-aspergillosis) prophylaxis.
  Interventions: Other: Patients without antifungal prophylaxis
- Patients with antifungal prophylaxis: Patients with acute myeloid leukemia treated with intensive chemotherapy. From 2012 to 2015, all patients received antifungal (anti-aspergillosis) prophylaxis by posaconazole.
  Interventions: Other: Patients without antifungal prophylaxis; Drug: Patients with antifungal prophylaxis

INTERVENTIONS:
Other: Patients without antifungal prophylaxis — Epidemiology data: clinical and biological informations collecting
Drug: Patients with antifungal prophylaxis — Hospitalized patients between 2012 and 2015 received Posaconazole prophylaxis during neutropenia period induced by induction or salvage chemotherapy.
  Groups: Patients with antifungal prophylaxis

SUMMARY:
Patients with acute myeloid leukemia (AML) are at risk to develop severe infections whose invasive aspergillosis (IA). These infections are leading to an important morbidity and mortality. Antifungal prophylaxis is recommended by posaconazole for AML patients during neutropenia induced by induction chemotherapy. Their application is not uniform.

DETAILED DESCRIPTION:
Invasive aspergillosis are frequent infections in hematological malignancy in particular during neutropenia induced by chemotherapy. Their incidence ranged between 5 to 25% according to the literature. Mortality may reach 30%. Our study described IA incidence in AML patients treated by intensive chemotherapy depending on antifungal prophylaxis by posaconazole. From 2009 to 2011, any patients received antifungal prophylaxis. From 2012 to 2015, patients received posaconazole during induction and salvage chemotherapy. During the all study period, efficacy of posaconazole is evaluated according to construction/demolition periods in hospital. All patients are hospitalized in High Efficiency Particulate Air (HEPA) filtration system.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* acute myeloid leukemia
* intensive chemotherapy (induction, consolidation, salvage, bone marrow transplantation)

Exclusion Criteria:

* < 18 years
* pregnancy
* no intensive chemotherapy (palliative treatment, azacytidine...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients treated for acute myeloid leukemia by intensive chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2009-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of invasive aspergillosis in acute myeloid leukemia | 1 year
  Evaluation of annual incidence of invasive aspergillosis in acute myeloid leukemia treated by intensive chemotherapy between 2009 and 2015

SECONDARY OUTCOMES:
Efficiency of antifungal prophylaxis by posaconazole | 1 year
  Comparison of two periods: 2009-2011 where patients had not antifungal prophylaxis and 2012-2015 where patients had antifungal prophylaxis by posaconazole during induction and salvage chemotherapy
Impact of antifungal prophylaxis by posaconazole about construction/demolition periods | 1 year
  Comparison of incidence of invasive aspergillosis while antifungal prophylaxis and construction/demolition periods

CONTACTS AND LOCATIONS:
Overall Officials: Gaelle Guillerm, MD, Principal Investigator — Department of Hematology, Brest Teaching Hospital; Lenaig Le Clech, MD, Principal Investigator — Department of Hematology, Brest Teaching Hospital
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No